CLINICAL TRIAL: NCT01201629
Title: Does Transcranial Direct Current Stimulation Improve Functional Motor Recovery in the Affected Arm-Hand in Patients After an Acute Ischemic Stroke: A Randomized Control Trial
Brief Title: Transcranial Direct Current Stimulation, Improve Functional Motor Recovery, Affected Arm
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual over 6 year period
Sponsor: University of Oklahoma (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1620
Record Dates: First submitted 2010-09-07; First posted 2010-09-14 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Brain Infarction; Brain Ischemia
Keywords: Ischemic Strokes; t DC stimulation; Functional recovery
MeSH Terms: conditions — Brain Infarction; Brain Ischemia; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- t DC stimulation (Sham Comparator): Sham transcranial direct current stimulation tDCS induces slight short-lasting tingling with onset of the stimulation. These sensations usually fade away in seconds. Sham interventions are essential to blind the subject and the assessor in order to obtain unbiased assessment of intervention effects
  Interventions: Device: t DC stimulation; Device: tDCStimulation
- tDC stimulation (Experimental): Actual DC stimulation
  Interventions: Device: t DC stimulation; Device: tDCStimulation

INTERVENTIONS:
Device: t DC stimulation — tDCS is a non-invasive, non-painful technique that modulates cortical excitability. tDCS can induce intracerebral current flow that is sufficiently large to achieve changes in cortical excitability. Thus, tDCS can be applied to humans non-invasively and painlessly to induce focal, lasting but reversible shifts of cortical excitability.
  Other Names: Sham transcranial DC brain stimulator
Device: tDCStimulation — 1 mA of tDCS will be delivered through surface electrodes (25-35 cm2) to the unaffected motor cortex for 30 min prior to a patient's scheduled OT. In the sham group patient will receive stimulation for 30 seconds only.
  Other Names: Experimental tDC stimulator

SUMMARY:
Overall goal of this study is to determine if transcranial direct current stimulation (tDCS) plus conventional occupational therapy improves functional motor recovery in the affected arm-hand in patients after an acute ischemic stroke compared to sham tDCS plus conventional occupational therapy, and to obtain information to plan a large randomized controlled trial.

DETAILED DESCRIPTION:
Study design:

Patients Successive admissions to the stroke service of the Veterans Affairs Medical Center with ischemic strokes will participate in this study.

Eligibility criteria:

Inclusion criteria:

1. Unilateral, 1st acute stroke event within 4 weeks of admission to an in-patient rehabilitation facility
2. Ischemic stroke documented clinically and by neuroimaging.
3. Severe upper limb weakness (MRC grade of 2 or less at the shoulder joint)
4. Medically stable from a cardio-respiratory stand point so that they can participate in daily therapies.
5. Depressed patients will be included in the study (psychiatrist referral will be made if deemed necessary).
6. Aphasic alert patients will be included in the study provided they were able to follow simple directions by verbal or gestural cues and provided with a written informed consent.
7. Informed consent, from cognitively intact patients (admission Mini Mental Scale Examination [MMSE] greater than or equal to 21). When it is not possible for the patient to provide informed consent or patient is cognitively impaired with MMSE ≤ 20, proxy consent will be obtained from the next of kin (legal authorized representative) according to institutional IRB standards. Informed consent will be obtained by the admitting physicians.

Exclusion criteria:

1. Hemorrhagic strokes
2. Patient's with an episode post-stroke seizure or history of epilepsy.
3. Patients medically unstable, demented, or terminally ill (e.g., patients with stroke as a complication of a terminal cancer).
4. On medications such as botox for spasticity or other medications known to enhance motor recovery such as d-amphetamine,
5. Stroke patients with implanted pacemakers and defibrillators.
6. Refusal to provide informed consent

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral, 1st acute stroke event within 4 weeks of admission to an in-patient rehabilitation facility
2. Ischemic stroke documented clinically and by neuroimaging.
3. Severe upper limb weakness (MRC grade of 2 or less at the shoulder joint)
4. Medically stable from a cardio-respiratory stand point so that they can participate in daily therapies.
5. Depressed patients will be included in the study (psychiatrist referral will be made if deemed necessary).
6. Aphasic alert patients will be included in the study provided they were able to follow simple directions by verbal or gestural cues and provided with a written informed consent.
7. Informed consent, from cognitively intact patients (admission Mini Mental Scale Examination [MMSE] greater than or equal to 21). When it is not possible for the patient to provide informed consent or patient is cognitively impaired with MMSE ≤ 20, proxy consent will be obtained from the next of kin (legal authorized representative) according to institutional IRB standards. Informed consent will be obtained by the admitting physicians.

Exclusion Criteria:

1. Hemorrhagic strokes
2. Patient's with an episode post-stroke seizure or history of epilepsy.
3. Patients medically unstable, demented, or terminally ill (e.g., patients with stroke as a complication of a terminal cancer).
4. On medications such as botox for spasticity or other medications known to enhance motor recovery such as d-amphetamine,
5. Stroke patients with implanted pacemakers and defibrillators.
6. Refusal to provide informed consent

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09-16 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meheroz H Rabadi, MD, MRCPI, Principal Investigator — Oklahoma University
Locations (1):
- Oklahoma City VA Medical Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2010 to 12/2015 at the OKC VA Med Center as in-patient
Pre-assignment Details: No significant events or enrolled participants were excluded.
Groups:
- Experimental (tDCs): t-DCs was administered in 8 patients externally for 30 min at 1 MA Anodal stimulation
- Sham: 8 patient received sham tDCs i.e. after 1 minute of tDCs the machine was off for the next 30 minutes.
Period: Overall Study
Arm/Group | Experimental (tDCs) | Sham
Started (Study started in 9/16/2010) | 8 | 8
Completed (Study terminated in 12/2015) | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental (tDCs) | Sham | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (11) | 63 (6) | 62 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1 | 3 | 4
  White | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Action Research Arm Test (ARAT) [Mean (Standard Deviation); unit: units on a scale] — Action Research Arm Test (ARAT), a standardized ordinal scale that measures UE function. 23 ARAT is based on the assumption that complex UE movements used in daily life can be explained and assessed by 4 basic movements: grasp, grip, pinch and gross movements of extension and flexion at the elbow and shoulder (Appendix 1). The ARAT is graded on a 4-point scale (0 is worse and 57 points is normal). ARAT scoring was undertaken as per instructions.
  units on a scale | 4 (10.9) | 1.9 (4.2) | 2.9 (8.1)
Functional Independence Measures (TFIM) [Mean (Standard Deviation); unit: units on a scale] — The FIM has 18 items and each item is scored on an ordinal scale ranging from 1 to 7. The total FIM score (TFIM) quantifies level of independence and ranges from 18 (total dependence) to 126 (total independence)
  units on a scale | 61 (17) | 59 (12) | 60 (14)

OUTCOME MEASURES:

1. Primary Outcome: Total Functional Independence Measure (TFIM) Change Scores
Description: The Functional Independence Measure (FIM™) will measure the degree of disability. The FIM scale is a reliable and valid functional assessment measure widely used in rehabilitation settings. The FIM has 18 items and each item is scored on an ordinal scale ranging from 1 to 7. A FIM™ item score of seven is categorized as "complete independence," while a score of one is "total assist" (patient performs less than 25% of task). The total FIM score (TFIM) quantifies level of independence and ranges from 18 (lowest) to 126 (highest) level of independence.
Time Frame: from baseline to 4-weeks of therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental (tDCs) | Sham
Number analyzed (Participants) | 8 | 8
units on a scale | 22.4 (15.7) | 25.3 (9.1)
Statistical Analysis 1: Comparison: Experimental (tDCs) vs Sham; Test type: Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Action Research Arm Test (ARAT) Change Scores
Description: The Action Research Arm Test (ARAT) is a standardized ordinal scale that measures upper extremity (arm and hand) function. This test assesses the ability to lift various sized objects to a height of 14.75 inches, move cylindrical shaped objects a distance of 14.75 inches, use pinch grasp to lift varying sized objects (such as a ball bearing, and a marble) between the thumb and the 3rd finger, and perform 3 gross upper extremity movements. Each upper extremity is evaluated individually. Score 0=no arm-hand movement and 57=normal
Time Frame: baseline to after 4-weeks of therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental (tDCs) | Sham
Number analyzed (Participants) | 8 | 8
units on a scale | 10.1 (13.5) | 1.7 (4.4)
Statistical Analysis 1: Comparison: Experimental (tDCs) vs Sham; Test type: Other; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Discharge Disposition
Description: Patient discharged home or to sub-acute facility
Time Frame: after 4 weeks of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental (tDCs) | Sham
Number analyzed (Participants) | 8 | 8
Participants
  Home | 4 | 3
  Subacute Facility | 4 | 5

ADVERSE EVENTS:
Time Frame: 3-months
Arm/Group | Experimental (tDCs) | Sham
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes